CLINICAL TRIAL: NCT01156688
Title: A Prospective Randomized Comparison Trial on the Use of Mifepristone With Sublingual or Buccal Misoprostol for Medical Abortions of Less Than 9 Weeks Gestation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Joyce Chai, University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HKCTR-1069
Record Dates: First submitted 2010-06-30; First posted 2010-07-05 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: Abortion, Legal
Keywords: medical abortion for pregnancy of less than 9 weeks gestation
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sublingual Misoprostol (Active Comparator)
  Interventions: Drug: Misoprostol
- Buccal misoprostol (Active Comparator)
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — sublingual 800mcg misoprostol 48 hours after oral 200mg mifepristone
  Arms: Sublingual Misoprostol
Drug: Misoprostol — buccal misoprostol 800mcg 48 hours after oral 200mg mifepristone
  Arms: Buccal misoprostol

SUMMARY:
The primary objective of this study is to compare the incidence of side effects of buccal and sublingual misoprostol when combined with mifepristone for medical abortions of less than 9 weeks gestation. The secondary outcome is to compare the complete abortion rate and induction-abortion interval between the two methods of administration of misoprostol.

DETAILED DESCRIPTION:
After mifepristone was approved by the United States Food and Drug Administration in 2000, the combination of mifepristone 200 mg and vaginal use of misoprostol 800 mcg became almost a standard of care in early medical abortion up to 63 days of gestation. When combined with mifepristone for medical abortion in the first trimester, vaginal administration of misoprostol is more effective, faster, and has a lower rate of ongoing pregnancy, and fewer gastrointestinal side effects than oral misoprostol.

Although misoprostol is more effective when given vaginally, most women prefer the oral route because this can avoid the uncomfortable vaginal examination and provide more privacy during medical induction. Another concern about vaginal administration is the potential risk of infection. In late March 2006, analyses of serious uterine infections following medical abortions by a regimen of oral mifepristone followed by vaginal misoprostol led Planned Parenthood Federation of America health centres to change the route of misoprostol administration. Given these concerns, alternative administration via sublingual (holding pills under the tongue) and buccal (holding pills in the cheek) routes have been investigated, as the misoprostol is absorbed directly and avoids the gastrointestinal system similar to vaginal administration.

A pharmacokinetic study showed that sublingual administration of misoprostol resulted in the greatest bioavailability when compared with oral or vaginal administration. In a randomized, cross-over pharmacokinetic study of 10 women by Schaff and colleagues of sublingual versus buccal misoprostol 800 mcg, the mean misoprostol plasma concentration-time curves at 4 hours and the maximum concentration were significantly higher for sublingual administration than the buccal route. However, buccal misoprostol administration resulted in fewer symptoms and was found to be more acceptable by women.

Buccal misoprostol 800 mcg after mifepristone 200 mg for terminating pregnancy through 63 days of gestation has a higher success rate and less ongoing pregnancy when compared with oral misoprostol, especially in pregnancies of 57-63 days. Adverse effect profiles were similar, although fever and chills were reported approximately 10% more often among women who took buccal misoprostol. When used for abortion through 56 days of gestation, buccal administration of misoprostol after mifepristone appears to be a highly effective and acceptable alternative compared with vaginal administration, and with similar adverse effects profile.

Medical abortions of less than 9 weeks gestation using sublingual misoprostol 800 mcg after mifepristone 200 mg has achieved complete abortion rate of 98.2% but is associated with more gastrointestinal side effects, fever, and chills when compared with vaginal route.

Both buccal and sublingual administration of misoprostol following mifepristone have been shown to be effective in inducing first trimester medical abortions, but with different side effects profile. No clinical trials have been conducted comparing buccal and sublingual administration of misoprostol in first trimester medical abortion. The purpose of the present study is to compare the incidence of side effects of buccal and sublingual misoprostol when combined with mifepristone.

ELIGIBILITY:
Inclusion Criteria:

* good general health
* older than the age of legal consent (i.e. >18 years old)
* requesting medical abortion and eligible for abortion
* on Day 1 of the study (day of mifepristone administration) the duration of pregnancy not more than 63 days as confirmed by pelvic ultrasound examination
* intrauterine pregnancy (intrauterine amniotic sac seen in US)
* willing to use other than hormonal or intra-uterine contraception until the first menses after termination of pregnancy
* if treatment fails she agrees to termination of pregnancy with the surgical method
* willing and able to participate after the study has been explained
* haemoglobin higher than 10g/L

Exclusion Criteria:

* a history or evidence of adrenal pathology, steroid-dependent cancer, porphyria, diastolic pressure over 95mm Hg, bronchial asthma, arterial hypotension.
* a history or evidence of thrombo-embolism, severe or recurrent liver disease or pruritus of pregnancy
* the regular use of prescription drugs before admission to the study
* the presence of an IUCD in utero
* breast-feeding
* multiple pregnancies
* heavy smokers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
to compare the incidence of side effects of buccal and sublingual misoprostol when combined with mifepristone for medical abortions of less than 9 weeks gestation. | within 43 days after mifepristone

SECONDARY OUTCOMES:
to compare the complete abortion rate | up to the time when patient's return of next mense, on average within 60 days after mifepristone
to compare the induction-abortion interval | from insertion of misoprostol to day of abortion process, within 15 days after mifepristone

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Chai, MBChB, Principal Investigator — The University of Hong Kong
Locations (1):
- Family Planning Association, Hong Kong, Hong Kong